CLINICAL TRIAL: NCT04889885
Title: Short Term Efficacy of High-intensity Laser Therapy to Alleviate Pain in Patients With Knee Osteoarthritis: a Double-blinded Randomized Controlled Trial
Brief Title: Short Term Efficacy of High-intensity Laser Therapy in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2016/242
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Knee Osteoarthritis
Keywords: High-intensity, pain, knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity laser therapy (HILT) (Experimental): The participants in the intervention group were treated by HILT which was applied to the knee joint (2-3 sessions a week for a total of 10 sessions) plus conservative treatment.
  Interventions: Device: High-intensity laser therapy (HILT)
- Sham laser (Sham Comparator): The control group received a sham laser by the same laser machine (2-3 sessions a week for a total of 10 sessions) plus conservative treatment.
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: High-intensity laser therapy (HILT) — HILT was done by Multiwave Locked System (MLS) laser therapy combining 2 laser wavelengths (808 and 905 nm) in order to strengthen the effects of HILT. The laser was applied on medial, lateral and posterior parts around the knee joint. The total energy per session was 562.5 Joules (J) which was done 2-3 times a week for a total of 10 sessions.
  Additionally, the participants received conservative treatment for knee OA such as education about the disease, proper activities, and exercise.
  Other Names: High-power laser therapy (HPLT)
  Arms: High-intensity laser therapy (HILT)
Device: Sham laser — The control group received a sham laser (2-3 times a week for a total of 10 sessions) plus conservative treatment as in the intervention group. The laser machine was the same as in the intervention group; however, the laser was applied without releasing laser energy to the knee joint.
  Arms: Sham laser

SUMMARY:
Knee osteoarthritis (KOA) is one of the most common health problems around the world. According to this, several interventions have been used to treat this group of patients including pharmacological and non-pharmacological management such as weight reduction, behavior modification, and physical therapy. Recently, high-intensity laser therapy (HILT) has been used to treat patients with KOA. The results of previous studies showed that HILT could help to reduce pain as well as improved function in patients with mild to moderate KOA. However, there were still no standardized guidelines for HILT treatment in KOA. Also, no previous studies evaluated the efficacy of HILT in patients with severe KOA. The present study, therefore, recruited not only mild to a moderate degree but also severe degree. The study aim was to determine the efficacy of HILT in terms of pain relief in patients with mild, moderate, and severe KOA. The hypothesis was HILT would effectively reduce pain in patients with KOA compared to sham laser plus conservative treatment.

DETAILED DESCRIPTION:
* This study is a double-blinded randomized control trial that compared the efficacy of HPLT to sham laser in patients with KOA.
* 42 patients who had KOA diagnosed by the American college of rheumatology (ACR) 2016 guidelines were recruited including a drop out of 20%.
* The participants were then randomly allocated into two groups (21 participants per group), mainly HILT and sham laser. Also, both groups received conservative treatment such as disease education, exercise, and advice for weight reduction.
* The intervention group received HILT which was applied on the medial, lateral, and posterior part of the knee joint. The total energy was 562.5 J per session which was done 2-3 sessions a week, for a total of 10 sessions.
* The control group received sham laser by the same device for 10 sessions plus conservative treatment as in the intervention group.
* The outcome measures, VAS and T-WOMAC score were recorded before and at the end of the study.
* Statistical analysis was performed using SPSS 18.0 version to evaluate the statistically significant change within the same group and the difference between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary knee OA diagnosed based on the American college of rheumatology (ACR) guidelines for early diagnosis of knee osteoarthritis 2016.
* Patients who had knee pain for at least 6 months and had VAS score greater than 4 out of 10 points
* Patients with knee OA who have Kellgren And Lawrence (KL) classification stages 2-4.

Exclusion Criteria:

* Patients who have secondary knee OA caused by other pathologies
* Patients who have a history of corticosteroid or hyaluronate injecting into the knee joint within the past 6 months
* Patients who were treated by physical therapy equipment within 1 month before the study
* History of stroke, bleeding disorders, cancer, deep vein thrombosis, cognitive impairment, or mental disorders
* Contraindicate to laser therapy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | VAS was recorded in the two time points. The first time point was at the baseline or before starting the treatment. After that, VAS was recorded post-intervention (at 4 weeks from baseline) as the second time point.
  VAS is the standardized pain measurement which allows subjects to rate pain score by using the ruler scale. This pain scale starts from 0 which means no pain to 10 which means maximum pain.

SECONDARY OUTCOMES:
Thai version of the Western Ontario and McMaster (WOMAC) Osteoarthritis Index for knee osteoarthritis (T-WOMAC) | T-WOMAC was recorded in the two time points. First, T-WOMAC was recorded at the baseline and was then recorded post-intervention (at 4 weeks from baseline) as the second time point.
  WOMAC score is the questionnaire used to assess pain and function in patients with knee OA. This score consists of 3 subscale including pain, function and joint stiffness. The total scores of all subscales are 96 points in which the higher score reflects the more disabled of the patient. For Thai version of WOMAC, this score has been proven valid for using in patients with knee OA.

REFERENCES:
- [Derived] Siriratna P, Ratanasutiranont C, Manissorn T, Santiniyom N, Chira-Adisai W. Short-Term Efficacy of High-Intensity Laser Therapy in Alleviating Pain in Patients with Knee Osteoarthritis: A Single-Blind Randomised Controlled Trial. Pain Res Manag. 2022 Oct 21;2022:1319165. doi: 10.1155/2022/1319165. eCollection 2022. PMID 36313402